CLINICAL TRIAL: NCT01332123
Title: Biomechanical Assessment of Gait in Lower-Extremity-Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Milwaukee (Other)
Responsible Party: Principal Investigator, Goeran Fiedler, Student-PI, University of Wisconsin, Milwaukee
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: UWM-11.254
Record Dates: First submitted 2011-04-06; First posted 2011-04-08 (Estimated); Results first posted 2016-06-09 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Prosthesis User

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alignment perturbations (Experimental): The following modifications will be applied to the prostheses: increased foot plantar flexion, increased foot dorsal flexion, increased foot supination, increased foot pronation (always 2 degrees from the neutral position)
  Interventions: Device: Alignment perturbations

INTERVENTIONS:
Device: Alignment perturbations — Increased foot plantar flexion, increased foot dorsal flexion, increased foot supination, increased foot pronation (always 2 degrees from the neutral position)

SUMMARY:
This study is investigating the influence of several simulated real life conditions on the symmetry of gait with trans-tibial prostheses

Hypotheses: It is hypothesized that the observable differences in gait pattern between amputees can be detected by a combination of forces and moments that are measured internally in the prosthesis, and electromyography data. It is further hypothesized that changing conditions such as uneven walking surface, prosthetic misalignment or user fatigue are characterized by typical values in the measured data or combinations thereof.

DETAILED DESCRIPTION:
In amputee walking, an optimal static alignment of the artificial leg is important in order to achieve the best possible performance. Comfort, energy expenditure, mobility and walking speed should ideally be similar to those of able bodied persons. Of course, amputation level, overall health status and other factors often pose certain individual limitations that may prevent an amputee from reaching this goal.

Irrespective of that, the artificial leg must be aligned properly to eliminate unnecessary inhibitions. Apart from manufacturing a well fitting socket, and selecting the appropriate functional components of the prosthesis, the prosthetist has to routinely optimize the static alignment during the fitting process. Hereby, objective measures and guidelines are scarce. Despite various more or less useful tools that are available, the alignment optimization in praxis is often based on subjective gait assessment and rules of thumb. Commonly accepted is the notion, that the gait pattern should be most symmetrically, that is step lengths, stance times, knee angles etc. should be identical between sound and prosthetic leg.

There are different questions that our study wants to address: Is gait symmetry indeed a valid measure of prosthetic performance (e.i. is it the most energy efficient way to walk)? How does the gait pattern change when the prosthesis user walks on different surfaces, becomes tired or tries to compensate for a less-than-optimal prosthesis fit? How can gait symmetry be objectively assessed without using an expensive motion analysis laboratory? We hope that our findings will provide practically useful information that can help improve prosthetic fittings in the field.

The study will be based on data from up to 15 trans-tibial prosthesis users. Participants will walk with their standard prosthesis, which will be equipped with a small sensor unit for the measurement of forces and moments during walking. The muscle activity of the thigh muscles will be measured using surface EMG sensors. All of the data collection will take place at the USR facilities (115 E Reindl Way, Milwaukee), where a multi camera motion analysis system is set up. Trials will require an overall time commitment of 5 hours at most, and will include normal walking, walking on carpet and gravel, walking up and down stairs, walking with fatigued thigh muscles.

ELIGIBILITY:
Inclusion Criteria:

* Trans tibial amputation
* Able to walk 30 minutes comfortably
* Modular prosthesis

Exclusion Criteria:

* Prosthesis does not provide enough space between socket and foot module to fit the mobile measuring unit
* Physically or mentally unable to perform the required tasks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-04; Primary Completion 2011-11 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brooke A Slavens, PhD, Principal Investigator — UWM CHS
Locations (1):
- USR, 115 E Reindl Way, Milwaukee, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Alignment Perturbations: The following modifications were applied to the prostheses: increased foot plantar flexion, increased foot dorsal flexion, increased foot supination, increased foot pronation, increased foot outward rotation, increased foot inward rotation (always 15 degrees from the neutral position)
  Alignment perturbations: Increased foot plantar flexion, increased foot dorsal flexion, increased foot supination, increased foot pronation, increased foot outward rotation, increased foot inward rotation (always 15 degrees from the neutral position)
Period: Overall Study
Arm/Group | Alignment Perturbations
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Alignment Perturbations
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (13.2)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Asymmetry Index
Description: Gait data was continuously recorded and was post processed to determine symmetry between left and right legs. Symmetry was computed by dividing the difference between legs by the average of both legs. 0 marks perfect symmetry and greater values higher asymmetry. There is no maximum limit.
  The overall asymmetry index was calculated as the mean of the following: max knee flex, dorsi flexion, plantar flexion (1st and 2nd peak), knee moment, dorsi-flexion moment, plantar-flexion moment, times of max in % of the gait cycle, Stance phase % of gait cycle and step length.
  The kinematics asymmetry index was calculated as the mean of the following: maximal knee flex, dorsi flexion, plantar flexion (1st and 2nd peak), the times of max in % of the gait cycle, Stance phase % of gait cycle and step length.
  The kinetics asymmetry index was calculated as the mean of the following variables: knee moment, dorsi-flexion moment, plantar-flexion moment, the times of max in % of the gait cycle.
Time Frame: 1 hour
Population: Two of the recruited participants were not included in the analysis, as they had bilateral amputations. Bilateral amputation was not posted as an exclusion criteria initially, but posted unanticipated limitations during data collection and analysis.
Measure: Mean (Standard Deviation); unit: unit-less index (0 = perfect symmetry)
Groups:
- Alignment Perturbations: The following modifications were applied to the prostheses: increased foot plantar flexion, increased foot dorsal flexion, increased foot supination, increased foot pronation (always 2 degrees from the neutral position)
  All participants were subjected to the same 5 interventions (neutral alignment and 4 perturbations as detailed above) in sequence to allow repeated measures (within-subject) comparisons.
Arm/Group | Alignment Perturbations
Number analyzed (Participants) | 8
unit-less index (0 = perfect symmetry)
  max knee flex | 0.064 (0.053)
  max dorsiflex | 0.352 (0.372)
  max plantarflex 1 | 0.541 (0.264)
  max pflex 2 | 1.481 (0.469)
  % time of max knee flex | 0.037 (0.025)
  % time of max dorsiflex | 0.111 (0.173)
  % time of pflex 1 | 0.238 (0.137)
  % time of pflex 2 | 0.038 (0.026)
  max knee moment | 0.792 (0.599)
  % time of max knee moment | 0.794 (0.589)
  max dflex moment | 0.137 (0.129)
  % time of max dflex moment | 0.178 (0.359)
  max pflex moment | 0.652 (0.598)
  % time of max pflex moment | 0.437 (0.556)
  stance phase % of cycle | 0.041 (0.026)
  step length | 0.076 (0.078)
  overall asymmetry index | 0.373 (0.124)
  kinematics asymmetry index | 0.298 (0.071)
  kinetics asymmetry index | 0.498 (0.339)

2. Secondary Outcome: Heart Rate Change
Description: Subjects were wearing a wireless heart rate monitor. The respective readings were noted and assessed during and immediately following the trials to estimate individual exertion rates. Changes in heart rate between resting and exertion across the sample were investigated to be able to interpret the primary outcome measures and to discuss limitations of the protocol. Unequal exertion rates within the sample would cause uneven trends biomechanical changes that are related to exertion.
Time Frame: 1 hour
Measure: Mean (Full Range); unit: beats/minute
Groups:
- Alignment Perturbations: The following modifications were applied to the prostheses: increased foot plantar flexion, increased foot dorsal flexion, increased foot supination, increased foot pronation (always 2 degrees from the neutral position)
  Alignment perturbations: Increased foot plantar flexion, increased foot dorsal flexion, increased foot supination, increased foot pronation (always 2 degrees from the neutral position)
Arm/Group | Alignment Perturbations
Number analyzed (Participants) | 8
beats/minute | 55.75 [31 to 78]

ADVERSE EVENTS:
Arm/Group | Alignment Perturbations
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 5/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alignment Perturbations (N=10)
Exertion (General disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes